CLINICAL TRIAL: NCT06973681
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase II Clinical Study to Evaluate the Safety, Tolerability, PK/PD Profile, and Efficacy of Multiple Doses of BGM0504 Injection in Overweight or Obese Subjects Without Diabetes
Brief Title: A Study of BGM0504 Evaluating Weight Loss in Overweight or Obese Chinese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGM0504-II-WL
Record Dates: First submitted 2025-05-14; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2023-06

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5 mg BGM0504 (Experimental): 5 milligrams (mg) BGM0504 administered subcutaneously (SC) once a week.
  Interventions: Drug: BGM0504
- 10 mg BGM0504 (Experimental): 10 mg BGM0504 administered SC once a week.
  Interventions: Drug: BGM0504
- 15 mg BGM0504 (Experimental): 15 mg BGM0504 administered SC once a week.
  Interventions: Drug: BGM0504
- Placebo (Placebo Comparator): Placebo administered SC once a week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGM0504 — Administered SC
  Arms: 10 mg BGM0504
Drug: BGM0504 — Administered SC
  Arms: 15 mg BGM0504
Drug: BGM0504 — Administered SC
  Arms: 5 mg BGM0504
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
To assess the effect of BGM0504 injection versus placebo on weight loss in overweight or obese subjects after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. BMI ≥ 28.0 kg/m2 or 24.0 ≤ BMI < 28.0 kg/m2 with at least 1 weight-related comorbidity at screening visit; 2.Controlled by diet and exercise alone for at least 12 weeks prior to Screening with <5.0% change in body weight and able to continue the original diet and exercise for weight control during the trial.

Exclusion Criteria:1.Those who have used weight loss drugs within 12 weeks before screening; 2. Previous diagnosis of type 1 or type 2 diabetes mellitus; 3. History of acute or chronic pancreatitis, or pancreatic injury; 4. History of thyroid C-cell carcinoma, MEN (multiple endocrine adenomatosis) 2A or 2B, or relevant family history; 5. Subjects with uncontrolled hypertension after treatment (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥ 100 mmHg at screening) or untreated blood pressure meeting the above criteria at screening; 6. Concomitant thyroid dysfunction that cannot be controlled at a stable drug dose atscreening, or clinically significant abnormalities in thyroid function test results at screening that require initiation of therapy; 7. At Screening, abdominal ultrasound indicated calculus gallbladder and polyps, or presence of clinical symptoms of gallbladder disease at Screening; 8. Pregnant or breastfeeding women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Percentage change in body weight | Week 0 to Week 24
  Percentage change from baseline in body weight after 24 weeks of treatment.

SECONDARY OUTCOMES:
Proportion of Subjects with weight loss of ≥5% | Week 0 to Week 24
  Proportion of Subjects with weight loss of ≥5% from baseline in body weight after 24 weeks of treatment
Change from baseline in waist circumference | Week 0 to Week 24
  Change from baseline in waist circumference after 24 weeks of treatment
Change from baseline in BMI | Week 0 to Week 24
  Change from baseline in BMI after 24 weeks of treatment
Change from baseline in fasting plasma glucose (FPG) | Week 0 to Week 24
  Change from baseline in fasting plasma glucose (FPG) after 24 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, China